CLINICAL TRIAL: NCT04662645
Title: Embedded Palliative Care in the Management of Advanced Thoracic Malignancies
Brief Title: Embedded Palliative Care in Managing Symptoms in Participants With Recurrent Stage III-IV Thoracic Malignancies and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Carolyn Presley, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-18116; NCI-2018-01209 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-06-26; First posted 2020-12-10 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Caregiver; Malignant Pleural Neoplasm; Metastatic Thymic Carcinoma; Recurrent Lung Carcinoma; Recurrent Thymic Carcinoma; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Thymoma; Lung Neoplasms | interventions — Palliative Care; Patient Comfort

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (embedded palliative care) (Experimental): Participants and caregivers undergo embedded palliative care comprising symptom management (physical and psychological), advanced directives and goals of care discussion, caregiver support, and referral for adjunctive supportive services as needed at each clinic visit.
  Interventions: Other: Palliative Therapy; Other: Questionnaire Administration

INTERVENTIONS:
Other: Palliative Therapy — Undergo embedded palliative care
  Other Names: Comfort Care; palliation; palliative care; Palliative Treatment; Symptom Management; Symptoms Management
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well embedded palliative care works in managing symptoms in participants with stage III-IV thoracic malignancies that has come back and their caregivers. Embedded palliative care may improve distress and anxiety in participants and caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine feasibility of embedding a palliative care (PC) physician within the James Thoracic Oncology Clinic.

II. To assess patient and caregiver outcomes over a 12-month period within an embedded onco-palliative care clinic model.

III. To evaluate and describe clinician attitudes and beliefs regarding utilization of embedded palliative care as well as symptoms of provider burnout.

IV. To analyze health care utilization among participants receiving embedded onco-palliative care.

OUTLINE:

Participants and caregivers undergo embedded palliative care comprising symptom management (physical and psychological), advanced directives and goals of care discussion, caregiver support, and referral for adjunctive supportive services as needed at each clinic visit.

After completion of study, patients are followed for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or metastatic cancer of the chest (lung, thymus, or pleura): stage III or IV, recurrent disease
* Patients will receive therapy (chemotherapy, immunotherapy, targeted therapy or radiation therapy) at The Ohio State University
* New patients (defined as patients who have received no therapy for metastatic disease or have started treatment for metastatic disease within the last 30 days) or established patients with advanced cancer receiving anti-cancer therapy, no limit on prior therapies
* Patient and caregiver must be able to read and understand consent form
* Patients must designate a willing caregiver to participate although caregiver consent is not required for patient participation

Exclusion Criteria:

* Patients who are already enrolled or have been previously enrolled in palliative care or hospice services as an outpatient. Inpatient palliative care consultation prior to enrollment is permitted
* Patients who do not qualify for active anti-cancer therapy and opt to enroll in hospice services prior to study enrollment
* Patients who are unable to read or understand consent form
* Patients receiving primary systemic treatment outside of Ohio State. Outside radiation therapy is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2020-12-05 (Actual)

PRIMARY OUTCOMES:
Acceptance from providers to assess utilization of palliative care services | Up to 12 months
  Acceptance will be evaluated utilizing provider surveys (to capture provider opinions on palliative care utilization) as well as rate of enrollment. Preliminary data will be summarized and collected. Confidence intervals will also be calculated for feasibility rates.
Demand of palliative care services to be evaluated | Up to 12 months
  Preliminary data will be summarized and collected. Confidence intervals will also be calculated for feasibility rates.
Capacity and productivity to be evaluated | Up to 12 months
  Clinician capacity and productivity will be evaluated by looking at scheduling as well as billing productivity. Preliminary data will be summarized and collected. Confidence intervals will also be calculated for feasibility rates.
Resource assessment of staff and space | Up to 12 months
  Resources required, including patient care rooms and nursing support will also be evaluated. Preliminary data will be summarized and collected. Confidence intervals will also be calculated for feasibility rates.
Symptom burden (patient outcome) supportive care screen | Up to 12 months
  Will be assessed using Supportive care screen.
Symptom burden (patient outcome) Functional Assessment of Cancer Therapy-Lung | Up to 12 months
  Will be assessed using Functional Assessment of Cancer Therapy-Lung
Symptom burden (patient outcome) using HADS | Up to 12 months
  Will be assessed using Hospital Anxiety and Depression Scale (HADS)
Symptom burden using National Comprehensive Cancer Network distress thermometer (patient outcome) | Up to 12 months
  Will be assessed using National Comprehensive Cancer Network distress thermometer
Anxiety assessment using Hospital Anxiety and Depression Scale (patient outcome) | Up to 12 months
  Anxiety assessed using the Hospital Anxiety and Depression Scale
Depression assessment using Hospital Anxiety and Depression Scale (patient outcome) | Up to 12 months
  Depression assessed using the Hospital Anxiety and Depression Scale
Functional status assessed using Functional Activities Scale (patient outcome) | Up to 12 months
  Functional status assessment using Functional Activities Scale (FAS)
Health care service needs assessed using Supportive Care Needs Survey Partners and Caregivers (SCNS- P and C) (Caregiver outcome) | Up to 12 months
  Caregiver needs assessment using Supportive Care Needs Survey - Patients & Caregivers (SCNC-P&C)
Psychological/emotional needs assessed using SCNS- P and C (Caregiver outcome) | Up to 12 months
  Caregiver needs assessment using Supportive Care Needs Survey - Patients & Caregivers (SCNC-P&C)
Work/social needs assessed using SCNS- P and C (Caregiver outcome) | Up to 12 months
  Caregiver needs assessment using Supportive Care Needs Survey - Patients & Caregivers (SCNC-P&C)
Information needs assessed using SCNS- P and C (Caregiver outcome) | Up to 12 months
  Caregiver needs assessment using Supportive Care Needs Survey - Patients & Caregivers (SCNC-P&C)
Self-reported barriers and attitudes regarding palliative care assessed using Ohio State Palliative Care Provider Survey (Provider outcome) | Up to 12 months
  Ohio State Palliative Care Provider survey used to assess perceived barriers to referral
Health care utilization outcomes | Up to 12 months
  Will be captured using Integrated Health Information Systems electronic medical record data as well as patient reported events.

SECONDARY OUTCOMES:
Challenges for patients, caregivers, and the treating oncologist in an embedded palliative care model | Up to 12 months
  evaluate the challenges for patients, caregivers and treating oncologist in embedded palliative care

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Presley, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT04662645/ICF_000.pdf